CLINICAL TRIAL: NCT02382640
Title: A Phase 1, Open-Label, Single Center, Single-Dose, Randomized, 4-Way Crossover Study to Assess the Effect of an Antacid on the Bioavailability of Febuxostat After Oral Administration of a 80 mg Febuxostat Extended-Release (XR) Capsule Formulation
Brief Title: Effect of Antacid on Bioavailability of Febuxostat After Administration of a Febuxostat 80 mg Extended-Release Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Febuxostat XR-1010; U1111-1163-1813 (Registry Identifier: WHO)
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1: ABDC (Experimental): Experimental: Sequence 1: ABDC Febuxostat 80 mg extended-release (XR) capsule, orally, once, after a 10-hour fast, and 20 mL Maalox Advance Regular Strength liquid containing Aluminum Hydroxide 200 mg, Magnesium Hydroxide 200 mg, and Simethicone 20 mg/5 mL (hereafter referred as Maalox) or equivalent, orally, once, after a 10-hour fast, on Day 1 of Period 1 (A), followed by a 7-day washout period, followed by Maalox or equivalent, orally, once, after a 9-hour fast, and febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast (1 hour after Maalox or equivalent), on Day 1 of Period 2 (B), followed by a 7-day washout period, followed by febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, on Day 1 of Period 3 (D), followed by a 7-day washout period, followed by febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after an 11-hour fast (1 hour after febuxostat), on Day 1 of Period 4 (C).
  Interventions: Drug: Febuxostat XR; Drug: Maalox Advance Regular Strength liquid
- Sequence 2: DACB (Experimental): Experimental: Sequence 2: DACB Febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, on Day 1 of Period 1, followed by a 7-day washout period, followed by febuxostat 80 mg extended-release (XR) capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after a 10-hour fast, on Day 1 of Period 2, followed by a 7-day washout period, followed by febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after an 11-hour fast (1 hour after febuxostat), on Day 1 of Period 3, followed by a 7-day washout period, followed by Maalox or equivalent, orally, once, after a 9-hour fast, and febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast (1 hour after Maalox or equivalent), on Day 1 of Period 4.
  Interventions: Drug: Febuxostat XR; Drug: Maalox Advance Regular Strength liquid
- Sequence 3: CDBA (Experimental): Febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after an 11-hour fast (1 hour after febuxostat), on Day 1 of Period 1, followed by a 7-day washout period, followed by febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, on Day 1 of Period 2, followed by a 7-day washout period, followed by Maalox or equivalent, orally, once, after a 9-hour fast, and febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast (1 hour after Maalox or equivalent), on Day 1 of Period 3, followed by a 7-day washout period, followed by Febuxostat 80 mg extended-release (XR) capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after a 10-hour fast, on Day 1 of Period 4.
  Interventions: Drug: Febuxostat XR; Drug: Maalox Advance Regular Strength liquid
- Sequence 4: BCAD (Experimental): Maalox or equivalent, orally, once, after a 9-hour fast, and febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast (1 hour after Maalox), on Day 1 of Period 1, followed by a 7-day washout period, followed by febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after an 11-hour fast (1 hour after febuxostat), on Day 1 of Period 2, followed by a 7-day washout period, followed by febuxostat 80 mg extended-release (XR) capsule, orally, once, after a 10-hour fast, and Maalox or equivalent, orally, once, after a 10-hour fast, on Day 1 of Period 3, followed by a 7-day washout period, followed by febuxostat 80 mg XR capsule, orally, once, after a 10-hour fast, on Day 1 of Period 4.
  Interventions: Drug: Febuxostat XR; Drug: Maalox Advance Regular Strength liquid

INTERVENTIONS:
Drug: Febuxostat XR — Febuxostat extended-release (XR) capsules
Drug: Maalox Advance Regular Strength liquid — Maalox Advance Regular Strength liquid containing Aluminum Hydroxide 200 mg, Magnesium Hydroxide 200 mg, and Simethicone 20 mg/5 mL or equivalent

SUMMARY:
The purpose of this study is to assess the effect of antacid administration, and its timing, on the bioavailability of a single dose of febuxostat extended-release (XR) 80 mg.

DETAILED DESCRIPTION:
The drug being tested in this study is called febuxostat extended-release (XR). Febuxostat XR is being tested to assess if antacids affect how the drug moves throughout the body. This study will look at lab safety and side effects in people who take febuxostat XR.

This cross-over study will enroll approximately 36 patients. Participants will be randomly assigned to one of four treatment sequences. All participants will receive the following study medications by the end of the study:

* Febuxostat XR 80 mg capsules
* Maalox Advance Regular Strength liquid containing Aluminum Hydroxide 200 mg, Magnesium Hydroxide 200 mg, and Simethicone 20 mg/5 mL or equivalent

All participants will be administered one dose of one or both of the study medications on Day 1 of four separate study periods.

This single-centre trial will be conducted in the United States. The overall time to participate in this study is up to 84 days. Participants will make 5 visits to the clinic including four 4-day periods of confinement to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult male or female aged 18 to 55 years, inclusive, by check-in (Day-1 of Period 1)
2. Weighs at least 50 kg (110 pounds), and has a body mass index (BMI) between 18.0 kg/m^2 to 30 kg/m^2, inclusive at Screening.
3. Has estimated glomerular filtration rate ≥90 mL/min

Exclusion Criteria:

Any participant who meets any of the following criteria will not qualify for entry into the study:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received febuxostat in a previous clinical study or as a therapeutic agent.
3. Has a known hypersensitivity to any xanthine oxidase inhibitor, xanthine compounds or any component of the formulation of febuxostat tablets (see Package Insert) or to caffeine.
4. Has a known hypersensitivity to aluminum, magnesium hydroxide, or any component of the formulation of antacid (Maalox Advanced Regular Strength or equivalent) (see Package Insert).
5. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
6. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [eg, cholecystectomy]).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United States from 23-Feb-15 to 04-May-15.
Pre-assignment Details: Healthy participants were enrolled in this 4 period cross over study to receive 4 regimens which included febuxostat extended release (XR) 80 milligram (mg) and Maalox suspension 20 milliliter (mL) based on different fasting conditions.
Groups:
- Regimen A, Then B, Then D, Then C: Regimen(Reg)A(Febuxostat XR 80mg,capsule, orally, single dose after a 10hour(hr) fast and concurrently with Maalox 20mL(200mg magnesium hydroxide, 200mg aluminum hydroxide, and 20mg simethicone/5mL)or equivalent brand antacid, suspension, orally, single dose) on Day1 of first intervention period(3 Days),followed by 1week washout period, followed by RegB(Maalox 20mL,suspension,orally, single dose after a 9hr fast,followed by Febuxostat XR 80mg,capsule, orally, single dose after a 10hr fast[or 1hr after antacid dose]) on Day1 of second intervention period(3Days),followed by 1 week washout period, followed by RegD(Febuxostat XR 80mg,capsule, orally, single dose after a 10hr fast) on Day 1 of third intervention period(3Days),followed by 1week washout period, followed by RegC(Febuxostat XR 80mg,capsule, orally, single dose after a 10hr fast followed by Maalox 20mL, suspension, orally, single dose after 11hr fast[or 1hr after Febuxostat dose]) on Day1 of fourth intervention period(3 Days).
- Regimen D, Then A, Then C, Then B: Regimen D (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast) on Day 1 of first intervention period (3 Days), followed by Regimen A (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast and concurrently with Maalox 20 mL, suspension, orally, single dose) on Day 1 of second intervention period (3 Days), followed by 1 week washout period, followed by Regimen C (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast followed by Maalox 20 mL, suspension, orally, single dose after 11-hour fast [or 1 hour after Febuxostat dose]) on Day 1 of third intervention period (3 Days), followed by 1 week washout period, followed by Regimen B (Maalox 20 mL, suspension, orally, single dose after a 9-hour fast, followed by Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast [or 1 hour after antacid dose]).
- Regimen C, Then D, Then B, Then A: Regimen C (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast followed by Maalox 20 mL, suspension, orally, single dose after 11-hour fast [or 1 hour after Febuxostat dose]) on Day 1 of first intervention period (3 Days), followed by 1 week washout period, Regimen D (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast) on Day 1 of second intervention period (3 Days), followed by 1 week washout period, Regimen B (Maalox 20 mL, suspension, orally, single dose after a 9-hour fast, followed by Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast [or 1 hour after antacid dose]) on Day 1 of third intervention period (3 Days), followed by Regimen A (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast and concurrently with Maalox 20 mL, suspension, orally, single dose) on Day 1 of fourth intervention period (3 Days).
- Regimen B, Then C, Then A, Then D: Regimen B (Maalox 20 mL, suspension, orally, single dose after a 9-hour fast, followed by Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast [or 1 hour after antacid dose]) on Day 1 of first intervention period (3 Days), followed by 1 week washout period, followed by Regimen C (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast followed by Maalox 20 mL, suspension, orally, single dose after 11-hour fast [or 1 hour after Febuxostat dose]) on Day 1 of second intervention period (3 Days), followed by Regimen A (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast and concurrently with Maalox 20 mL, suspension, orally, single dose) on Day 1 of third intervention period (3 Days), Regimen D (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast) on Day 1 of fourth intervention period (3 Days).
Period: Intervention Period 1 (3 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 2 (3 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 3 (3 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 4 (3 Days)
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D
Started | 9 | 9 | 9 | 9
Completed | 8 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Laboratory Abnormality | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set was defined as all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A, Then B, Then D, Then C | Regimen D, Then A, Then C, Then B | Regimen C, Then D, Then B, Then A | Regimen B, Then C, Then A, Then D | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (7.36) | 34.7 (13.42) | 31.7 (9.18) | 35.8 (11.38) | 35.0 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 6 | 21
  Male | 4 | 4 | 4 | 3 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 3 | 4 | 5 | 17
  Not Hispanic or Latino | 4 | 6 | 5 | 4 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 2 | 4 | 3 | 10
  White | 8 | 6 | 5 | 5 | 24
  Multiracial | 0 | 1 | 0 | 1 | 2
Smoking classification [Number; unit: participants]
  Has never smoked | 8 | 9 | 8 | 8 | 33
  Is an ex-smoker | 1 | 0 | 1 | 1 | 3
Alcohol classification [Number; unit: participants]
  Has never drunk | 2 | 4 | 5 | 4 | 15
  Is a current drinker | 4 | 1 | 1 | 2 | 8
  Is an ex-drinker | 3 | 4 | 3 | 3 | 13
Xanthine/caffeine consumption [Number; unit: participants]
  Had xanthine/caffeine consumption | 5 | 5 | 3 | 5 | 18
  Had no xanthine/caffeine consumption | 4 | 4 | 6 | 4 | 18
Female reproductive status [Number; unit: participants]
  Female of childbearing potential | 4 | 5 | 4 | 4 | 17
  Surgically sterile | 1 | 0 | 1 | 2 | 4
  N/A (participant is male) | 4 | 4 | 4 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Febuxostat
Time Frame: Days 1 at multiple timepoints (up to 48 hours) post-dose
Population: The pharmacokinetic set consisted of all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Regimen A: Regimen A (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast and concurrently with Maalox 20 mL, suspension, orally, single dose) on Day 1 in either of the 4 intervention periods
- Regimen B: Regimen B (Maalox 20 mL, suspension, orally, single dose after a 9-hour fast, followed by Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast [or 1 hour after antacid dose]) on Day 1 in either of the 4 intervention periods.
- Regimen C: Regimen C (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast followed by Maalox 20 mL, suspension, orally, single dose after 11-hour fast [or 1 hour after Febuxostat dose]) on Day 1 in either of the 4 intervention periods.
- Regimen D: Regimen D (Febuxostat XR 80 mg, capsule, orally, single dose after a 10-hour fast) on Day 1 in either of the 4 intervention periods.
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
nanogram per milliliter (ng/mL) | 883.58 (898.49) | 1075.08 (941.46) | 765.89 (480.2) | 1456.42 (875.39)

2. Primary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve During the Dosing Interval for Febuxostat
Time Frame: Days 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
nanogram*hour per milliliter (ng*hr/mL) | 4680.69 (2427.11) | 5877.99 (2888.9) | 4412.22 (1718.42) | 7316.21 (2811.1)

3. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Febuxostat
Time Frame: Days 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
ng*hr/mL | 5901 (2739.92) | 6999.9 (2912.71) | 4844.33 (1918.73) | 7697.85 (2732.63)

4. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to 30 days after last dose of drug (Day 31 for each of the 4 periods)
Population: The safety set was defined as all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
participants
  TEAE | 2 | 1 | 3 | 2
  SAE | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Day 1 up to 30 days after last dose of drug (Day 31 for each of the 4 periods)
Population: The safety set was defined as all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
participants | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings
Time Frame: Day 1 up to 30 days after last dose of drug (Day 31 for each of the 4 periods)
Population: The safety set was defined as all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Evaluation
Time Frame: Day 1 up to 30 days after last dose of drug (Day 31 for each of the 4 periods)
Population: The safety set was defined as all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
participants | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG)
Time Frame: Day 1 up to 30 days after last dose of drug (Day 31 for each of the 4 periods)
Population: The safety set was defined as all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 36 | 36 | 35 | 36
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 2/36 | 1/36 | 3/35 | 2/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (N=36) | Regimen B (N=36) | Regimen C (N=35) | Regimen D (N=36)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral herpes (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.